## Summary of protocol for post-marketing surveillance (031-101-00116)

## - Aripiprazole for irritability associated with pediatric autism spectrum disorder (ASD) in Japan

| Study Title | Abilify special-drug-use-results survey (pediatric autism spectrum disorder: oral |
|---|---|
| | formulations) |
| Study Code | 031-101-00116 |
| Name of Company | Otsuka Pharmaceutical Co., Ltd. |
| Responsible party | Office of Surveillance Management, Pharmacovigilance Department |
| Product Name | ABILIFY Tablets(Aripiprazole), ABILIFY Powder(Aripiprazole), ABILIFY Oral |
| | Solution(Aripiprazole), ABILIFY OD Tablets (Aripiprazole) |
| Product, Dose | Drug products investigated: |
| | ABILIFY Tablets 1mg / 3mg /6mg /12mg |
| | ABILIFY Powder 1% |
| | ABILIFY Oral Solution 0.1% |
| | ABILIFY OD Tablets 3mg /6mg /12mg |
| | Dosage and Administration: |
| | The usual starting dose in children (from 6 to 17 years old) is 1 mg of |
| | aripiprazole per day administered. Maintenance dose are from 1mg to 15 mg per |
| | day are administrated. The dose may be changed for symptom, The fluctuation of |
| | dose are restricted to 3mg per day. |
| Clinical Phase | IV (non-interventional study) |
| Rationale and | Observational study conducted in Japan is based on the re-examination system and |
| background | not as a condition of the marketing authorization. This kind of non-interventional |
| | study is generally imposed to all new drugs to quantify the incidence of adverse |
| | drug reactions (ADRs), and not requested to identify the safety concerns. |
| | The re-examination system in Japan is defined by the article 14-4 of the |
| | Pharmaceutical Affairs Law. During a period of re-examination, the MAH plans |
| | and conducts post-marketing surveys based on GPSP ordinance. In meantime, |
| | results from post-marketing surveys are reported periodically to PMDA based on |
| | Periodic Safety Reports (Article 63 of the Enforcement Regulations of the Law). |
| Objective | The purpose of this survey is to identify the following safety and efficacy-related |
| | questions for an observation period of 1 year with use of oral drug of Abilify in the |
| | routine clinical setting. |
| Study design | Observational study |
| | (Multicenter, prospective post-marketing surveillance) |
| Data source | Not applicable (Primary data collection) |
| [ | 1 |

| Population | Pediatric patients in Japan with irritability associated with autism spectrum disorder |
|---|---|
| | who are planned to be newly started on oral drug of Abilify. |
| Sample size | 300 patients |
| Study Period | Study period: April 2017 to September 2019 (30 months) |
| | Enrollment period: April 2017 to June 2018 (15 months) |
| | End of Data collection: December 2019 |
| Primary end point | For each patient, the observation period is 1 year from the start date of oral drug of |
| | Abilify. |
| | For patients who discontinue oral drug of Abilify therapy within 1 year, the |
| | observation period is to be up to the date of discontinuation of Abilify |
| | administration. |
| Methodology | Safety information is collected with the procedure described in applicable SOPs. |
| | Safety Information is defined as "Any information from any source containing |
| | information such as: |
| | Adverse event or suspicion thereof |
| | • Lack of efficacy |
| | Overdose/incorrect dosage (accidental or intentional) |
| | • Abuse/misuse (e.g. patients sharing medication) – even without resulting adverse |
| | reaction |
| | Accidental exposure (e.g. child takes parent's medication) |
| | Medication error |
| | Withdrawal reactions |
| | Disease progression/exacerbation of existing disease |
| | Drug-drug/Drug-food interactions |
| | • Exposure to drug during pregnancy, where the embryo or fetus may have been |
| | exposed to medicinal products (either through maternal exposure or transmission |
| | of a medicinal product via semen following paternal exposure). |
| | Exposure to drug during lactation (including uneventful) |
| | Suspected counterfeit product |
| | • Suspected transfer of infectious disease/agent by the medicinal product concerned. |
| | · Product Quality Complaint (PQC) with safety related/medically important |
| | information |
| | Pediatric use (if not an approved use) |
| | Occupational exposure |
| | • Off-label use |
| | Data entry system for original data: PostMaNet (Ver.4) (an electronic data |

| | capturing system of Fujitsu FIP Corporation) |
|---|---|
| | Forwards Safety Information from any source to the Local Safety Manager (LSM) |
| | or appropriate local PV Representative within 24 hours of awareness or the next |
| | working day in the case of receipt the day prior to or during a weekend, but no later |
| | than 3 calendar days for reporting to the Global Case Receipt Mailbox. |
| | Type of CRF: eCRF |
| Reconciliation | The reconciliation of the serious and non-serious AEs between PV database (Argus) |
| | and study database is going to be performed on a monthly basis and at the end of the |
| | study. |
| Final study report | The FSR will be finalized within one year of the end of data collection |
| | (30 December 2020). |